CLINICAL TRIAL: NCT05722327
Title: Phase I Trial of Adagrasib (MRTX849) in Combination With Cetuximab and Irinotecan in Patients With Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mirati Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0374; NCI-2023-01157 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — adagrasib; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1 ( MRTX849 and Irinotecan) (Experimental): Participants assigned to Stage 1, participants dose levels of MRTX849 and irinotecan will depend on when the participants joined the study. This study will also test 2 different dosing schedules: concurrent dosing or staggered dosing
  Interventions: Drug: MRTX849; Drug: Irinotecan; Drug: Cetuximab
- Stage 2 ( MRTX849 and Irinotecan) (Experimental): Participants assigned to Stage 2 will receive MRTX849 and irinotecan at the dose level that was recommended during Stage 1. This study will also test 2 different dosing schedules: concurrent dosing or staggered dosing
  Interventions: Drug: MRTX849; Drug: Irinotecan; Drug: Cetuximab

INTERVENTIONS:
Drug: MRTX849 — Given by PO (mouth)
Drug: Irinotecan — Given by IV (vein)
Drug: Cetuximab — Given by IV (vein)
  Other Names: C225; Erbitux™; MC-C225; MOAB C225

SUMMARY:
To find the recommended dose of MRTX849 that can be given in combination with cetuximab and irinotecan to patients with colorectal cancer that have a mutation (genetic change) called KRAS G12C.

DETAILED DESCRIPTION:
Primary objectives:

* To determine the optimal biological dose (OBD) of MRTX849 when used in combination with cetuximab and irinotecan.
* To evaluate the safety profile of this combination.
* To determine the antitumor activity of this combination in patients with metastatic KRASG12C colorectal cancer.

Exploratory objectives:

* To explore correlations between MRTX849 exposure and patient outcomes such as disease response, objective response rate (ORR), duration or response (DOR), progression-free survival (PFS), overall survival (OS), safety, and pharmacodynamic endpoints.
* To evaluate the utility of detecting KRASG12C mutation in plasma to identify suitable patients.
* To explore potential pharmacodynamic (PD) markers of KRASG12C and EGFR inhibition in tumor tissue and/or blood plasma.
* To explore correlations between baseline tumor biomarkers, gene alterations, and clinical activity/efficacy.
* To define mechanisms of acquired resistance to EGFR and KRASG12C inhibition and evaluate novel strategies to overcome such resistance.
* To assess pharmacokinetics of MRTX849 and irinotecan and key metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the colon or rectum with KRASG12C mutation. KRASG12C on ctDNA may also be used as basis of eligibility, with approval from study or site PIs.
* Unresectable or metastatic disease.
* Previously treated with at least two prior chemotherapy regimens for metastatic disease (where a regimen is defined as a unique combination of 5-FU, oxaliplatin, irinotecan, bevacizumab (or biosimilar), capecitabine). A treatment with adjuvant therapy with progression within 6 months of completing therapy would be considered a prior chemotherapy regimen.
* Presence of tumor lesions to be evaluated per RECIST 1.1patients must have measurable disease.
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of the proposed combination in patients <18 years of age, and because solid tumor malignancies with KRASG12C mutation is rare among patients < 18 years of age, children are excluded from this study.
* Able to take oral medications.
* Most recent prior systemic therapy (e.g., chemotherapy, immunotherapy or, investigational agent) and radiation therapy discontinued at least 2 weeks before first dose or five half-lives whichever is shorter.
* Recovery from the adverse effects of prior therapy at the time of enrollment to ≤ Grade 1 (excluding alopecia and prior oxaliplatin-induced neuropathy).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Laboratory values within the screening period:

  * Absolute neutrophil count ≥ 1,000/mm3 (≥ 1.0, 109/L)
  * Platelet count ≥ 100,000/mm3 (≥ 100, 109/L)
  * INR/PTT ≤ 1.5 upper limit of normal (ULN)
  * Hemoglobin ≥ 9 g/dL, in the absence of transfusions for at least 2 weeks
  * Total bilirubin ≤ 1.5 upper limit of normal (ULN) (if associated with Gilbert's disease or UGT1A1*28 homozygosity, ≤ 3 ULN)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 ULN (if associated with liver metastases ≤5 ULN)
  * Estimated creatinine clearance ≥ 60 mL/min by Cockcroft-Gault or CKD-EPI.
* Women of child-bearing potential or men whose partner is a woman of child-bearing potential agree to use contraception while participating in this study, and for 6 months following termination of study treatment.
* Completed informed consent process, including signing of IRB-approved informed consent form.
* Willing and able to comply with clinical trial instructions and requirements.

Exclusion criteria:

* Active brain metastases, unless adequately treated and patient is neurologically stable (except for residual symptoms of central nervous system treatment) for at least 2 weeks prior to enrollment without corticosteroids or are on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent).
* Prior treatment with KRASG12C inhibitor + EGFR inhibitor combo
* Patients with carcinomatous meningitis.
* History of significant hemoptysis or hemorrhage within 4 weeks of the first dose, unless resolved or stable.
* Major surgery within 4 weeks of first dose.
* History of intestinal disease or major gastric surgery likely to alter absorption of study treatment.
* Any of the following cardiac abnormalities:

  * Symptomatic or uncontrolled atrial fibrillation or other arrhythmia
  * Unstable angina pectoris or myocardial infarction within the last 6 months.
  * Congestive heart failure ≥ NYHA Class 3 within the last 6 months.
  * QTc > 480 milliseconds.
  * LVEF, if known, beyond the allowable window for single-agent MRTX849
* Ongoing need for a medication with any of the following characteristics that cannot be switched to alternative treatment prior to study entry (see Appendix 2): known risk of Torsades de Pointes or QT prolongation; substrate of CYP3A with narrow therapeutic index; strong inducer or inhibitor of CYP3A and/or P-gp; strong inhibitor of BCRP; and proton pump inhibitors.
* Known or suspected presence of another malignancy that could be mistaken for the malignancy under study.
* Known human immunodeficiency virus (HIV) seropositivity or active Hepatitis B or C. Patients treated for hepatitis C with no detectable viral load are permitted.
* Pregnancy. Women of child-bearing potential must have a negative serum or urine pregnancy test during screening.
* Breast-feeding or planning to breast feed during the study or within 6 months after end of treatment.
* Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org